CLINICAL TRIAL: NCT05787171
Title: A Prospective Study to Compare the Cosmetic Results of Sutures With Different Absorption Rates for Lower Abdominal Incision
Brief Title: Three Sutures With Different Absorption Rates for Lower Abdominal Incision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJTU1AF2021CRF-019
Record Dates: First submitted 2022-08-25; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2022-10

CONDITIONS: Cicatrix
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PDS group (Experimental): The skin around the incision is dissociated from the bottom, followed by measuring the length of the wound and dividing it into three segments evenly. Each segment randomly received 2-0 Vicryl suture, 2-0 PDS suture, or 2-0 Ethibond suture to sew up the incision with WE-MBVMS. This is the group which received 2-0 PDS suture to sew up the incision.
  Interventions: Device: WE-MBVMS using suture PDS (polydioxanone; Johnson & Johnson International, USA)
- Vicryl group (Experimental): The skin around the incision is dissociated from the bottom, followed by measuring the length of the wound and dividing it into three segments evenly. Each segment randomly received 2-0 Vicryl suture, 2-0 PDS suture, or 2-0 Ethibond suture to sew up the incision with WE-MBVMS.This is the group which received 2-0 Vicryl suture to sew up the incision.
  Interventions: Device: WE-MBVMS using suture Vicryl (Polyglactin 910; Johnson & Johnson International, USA);
- Ethibond group (Experimental): The skin around the incision is dissociated from the bottom, followed by measuring the length of the wound and dividing it into three segments evenly. Each segment randomly received 2-0 Vicryl suture, 2-0 PDS suture, or 2-0 Ethibond suture to sew up the incision with WE-MBVMS.This is the group which received 2-0 Ethibond suture to sew up the incision.
  Interventions: Device: WE-MBVMS using suture Ethibond (polyester; Johnson & Johnson International, USA）

INTERVENTIONS:
Device: WE-MBVMS using suture Vicryl (Polyglactin 910; Johnson & Johnson International, USA); — The skin around the incision is dissociated from the bottom, followed by measuring the length of the wound and dividing it into three segments evenly. Each segment randomly received 2-0 Vicryl suture, 2-0 PDS suture, or 2-0 Ethibond suture to sew up the incision with WE-MBVMS.
  Arms: Vicryl group
Device: WE-MBVMS using suture PDS (polydioxanone; Johnson & Johnson International, USA) — The skin around the incision is dissociated from the bottom, followed by measuring the length of the wound and dividing it into three segments evenly. Each segment randomly received 2-0 Vicryl suture, 2-0 PDS suture, or 2-0 Ethibond suture to sew up the incision with WE-MBVMS.
  Arms: PDS group
Device: WE-MBVMS using suture Ethibond (polyester; Johnson & Johnson International, USA） — The skin around the incision is dissociated from the bottom, followed by measuring the length of the wound and dividing it into three segments evenly. Each segment randomly received 2-0 Vicryl suture, 2-0 PDS suture, or 2-0 Ethibond suture to sew up the incision with WE-MBVMS.
  Arms: Ethibond group

SUMMARY:
The previous studies have demonstrated that wedge excision combined modified buried vertical mattress suture (WE-MBVMS) provides better aesthetic outcomes than traditional ways. Prolonged tension reduction is crucial in WE-MBVMS suppressing scar, while suture used during WE-MBVMS decided the length of tension reducing time to a certain degree. However, presently surgeons select suture for WE-MBVMS mostly according to their personal preference and clinical experience and clinical comparative evidence exposing the best suture for desired cosmetic outcome is lacking. Here, investigators purposed to establish a feasibility trial comparing the scars left by WE-MBVMS using sutures with different tension holding time.

This is a feasibility, single-center RCT with 35 patients aiming to compare the scar of the hypogastric incision sutured by three different-absorption-rate sutures with WE-MBVMS. The incision induced by donating skin grafts is evenly divided into three segments, each segment randomly uses one of three different sutures randomly allocated by the SAS (V.9.4) statistical software. The feasibility of this study will be assessed by the primary outcomes, including patient and clinician enrolment refusal as well as their reasons, reasons for ineligibility, recruitment ratio, retention and withdrawal at each follow-up point (1, 3, and 6 months), reasons for withdrawal, integrity of collected data and adverse event rates. Secondary outcome measures of the cosmetic outcome of scar will help shape future fully powered RCT by formulating the sample size.

DETAILED DESCRIPTION:
Data from clinical trial and the previous study have demonstrated that wedge excision combined modified buried vertical mattress suture (WE-MBVMS) provides better aesthetic outcomes than traditional ways. As an effectively tension reducing, precisely edge everting and easily performing technique, WE-MBVMS has the following characteristics distinguishing it from other methods: (1) The edge of the incision was excised in a wedge size to guarantee a fully eversion in the edges of the incision; (2) And the stitch embed in the dermis as long as possible to recruit dermal tissue as much as possible in the suture loop, from which a sufficient skin eversion accompanied with visible skin folds is formed.

After the above operation, tension of the incision is effectively reduced and reserved to antagonist the consistently existing tension for a certain time, which is the core of WE-MBVMS in inducing slight scars. Although WE-MBVMS possesses the ability of confronting tension for a long time, the absorbable suture used during the WE-MBVMS decided the length of the tension reserving time. It is known that the period of scar molding is as long as 6-12 months, during which tension reducing contributes a lot in scar suppression. Hence, selecting appropriate material for the WE-MBVMS to achieve enough support for tension reducing of the incision might consequently lead to ideal scar suppression.

Nowadays, various kinds of absorbable sutures can be used in intradermal suture, among which PDS™ (polydioxanone) and Vicryl™ (polyglactin) is most commonly used. With the tension holding time of 90 days and 30 days, respectively, it is easy to relate them to different scar suppressing ability. Considering the crucial role of reducing tension played in suppressing scar and that nonabsorbable suture, also used in intradermal suture, provide prolonged dermal support, the researchers also employed polyester nonabsorbable suture in the WE-MBVMS . Although the ability of polyester suture in reducing tension will not be disturbed by its broken down by the body, tissue cutting and displacement will happen under the continuous action of external force over time. It follows that the efficiency of tension reduction and tissue eversion brought by polyester is prolonged but not permanent.

In this study, the lower abdominal incision will be selected which induced by harvesting autogenous skin grafts for wound repair to perform the comparison of the above three sutures. Because the donation causes incision, which leaves scar in the donor site that is mostly neglected by surgeons but concerned by patients. Besides, the hypogastrium is one of the important aesthetic units, thus scar is aesthetically undesirable or symptomatic8. Moreover, autogenous hypogastric skin graft, as an important skin donor site, is commonly used by plastic surgeons. Through comparing the cosmetic results of scars achieved by materials with different tension holding time, the researchers will further understand the duration of tension-reduction required for optimal scar inhibition and get a reference for suture selection. Taken together, a feasibility trial is required to produce more evidence for a fully powered randomised controlled trial (RCT).

This is a feasibility, single-center RCT with 35 patients aiming to compare the scar of the hypogastric incision sutured by three different-absorption-rate sutures with WE-MBVMS. The incision induced by donating skin grafts is evenly divided into three segments, each segment randomly uses one of three different sutures randomly allocated by the SAS (V.9.4) statistical software. The feasibility of this study will be assessed by the primary outcomes, including patient and clinician enrolment refusal as well as their reasons, reasons for ineligibility, recruitment ratio, retention and withdrawal at each follow-up point (1, 3, and 6 months), reasons for withdrawal, integrity of collected data and adverse event rates. Secondary outcome measures of the cosmetic outcome of scar will help shape future fully powered RCT by formulating the sample size.

ELIGIBILITY:
Inclusion Criteria:

* surgical incisions need to be closed after skin gotten;
* incisions at least 10 cm in length;
* patients aged between18 and 60 years old.

Exclusion Criteria:

* chronic diseases, like diabetes, chronic kidney disease, malignant neoplasms and severe malnutrition;
* pregnancy;
* inability to return for the follow-up visit;
* unwillingness to provide informed consent;
* inability to read or speak Chinese.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 1 month after the surgery
  As a 10cm line with 0 presenting the worst and 10 presenting the best overall satisfaction, the score of VAS is collected by patients placing a vertical mark on the VAS.
Visual Analogue Scale (VAS) | 3 month after the surgery
  As a 10cm line with 0 presenting the worst and 10 presenting the best overall satisfaction, the score of VAS is collected by patients placing a vertical mark on the VAS.
Visual Analogue Scale (VAS) | 6 month after the surgery
  As a 10cm line with 0 presenting the worst and 10 presenting the best overall satisfaction, the score of VAS is collected by patients placing a vertical mark on the VAS.
Patient Scar Assessment Scale (PSAS) | 1 month after the surgery
  Six domains including pain, itching, colour, pliability, thickness and relief, are contained in the PSAS.
Patient Scar Assessment Scale (PSAS) | 3 month after the surgery
  Six domains including pain, itching, colour, pliability, thickness and relief, are contained in the PSAS.
Patient Scar Assessment Scale (PSAS) | 6 month after the surgery
  Six domains including pain, itching, colour, pliability, thickness and relief, are contained in the PSAS.
Observer Scar Assessment Scale (OSAS) | 1 month after the surgery
  Six domains including pain, itching, colour, pliability, thickness and relief, are contained in the OSAS.
Observer Scar Assessment Scale (OSAS) | 3 month after the surgery
  Six domains including pain, itching, colour, pliability, thickness and relief, are contained in the OSAS.
Observer Scar Assessment Scale (OSAS) | 6 month after the surgery
  Six domains including pain, itching, colour, pliability, thickness and relief, are contained in the OSAS.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No